CLINICAL TRIAL: NCT03329937
Title: An Open-Label, Single-arm Pilot Study Evaluating the Antitumor Activity and Safety of Niraparib as Neoadjuvant Treatment in Localized, HER2-negative, BRCA-mutant Breast Cancer Patients
Brief Title: Study Evaluating the Antitumor Activity and Safety of Niraparib as Neoadjuvant Treatment in Participants With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213355; 3000-01-005 (Other: Tesaro)
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms, Breast
Keywords: Niraparib; Human epidermal growth factor receptor; Breast cancer; Breast ultrasound; Magnetic resonance imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with HER2-negative and BRCAmut breast cancer (Experimental): Participants with HER2-negative and BRCAmut localized breast cancer (primary tumor >=1 cm) will receive niraparib (200 mg PO).
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib is a potent, orally active, highly selective poly adenosine diphosphate ([ADP]-ribose) polymerase 1 (PARP1) and PARP2 inhibitor. It will be supplied as 100 mg capsules and will be administered at starting dose of 200 mg PO daily throughout 28 days for 2 cycles (each cycle is 28 days), with the potential for an additional 4 cycles (maximum total of 6 cycles) at the assigned dose and schedule.

SUMMARY:
This is an open-label, single-arm pilot study evaluating the antitumor activity and safety of niraparib as neoadjuvant therapy in participants with Human epidermal growth factor receptor 2 (HER2)-negative and breast cancer susceptibility gene mutant (BRCAmut) localized breast cancer (primary tumor >=1 centimeters [cm]). Breast magnetic resonance imaging (MRI), breast ultrasound, and tumor core biopsy will be performed at the screening (Days -28 to -1). Participants will receive niraparib (200 milligrams [mg] orally [PO]) treatment daily for 28 days (Cycle 1) and then will undergo breast ultrasound at the end of Cycle 1 on Day 28. Based on breast ultrasound reports, the participants will either discontinue the study (disease progression) or will continue niraparib treatment (complete response [CR], partial response [PR] or stable disease [SD]) for an additional cycle (Cycle 2). A breast MRI and breast ultrasound will be performed at the end of Cycle 2. Approximately 21 participants will be enrolled in this study and the study duration will be approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants age >= 18 years old.
* Participants with a deleterious or suspected deleterious breast cancer susceptibility gene 1 (BRCA1) or BRCA2 mutation (germline or somatic) may be enrolled into the study based on either local or central laboratory testing of BRCA status.
* Histologically-confirmed HER2-negative localized breast cancer by core biopsy.
* Primary operable, non-metastatic invasive carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration is not sufficient. Incisional biopsy is not allowed. In participants with multifocal and/or multicentric, the largest lesion should be measured. Both unilateral and bilateral breast cancer are allowed.
* Primary tumor size >=1cm.
* Measurable disease by breast ultrasound and MRI.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function defined as:

  1. Absolute neutrophil count (ANC) >=1500 per microliters (/μL).
  2. Platelets >=100,000/μL.
  3. Hemoglobin >=9 grams per deciliter (g/dL).
  4. Serum creatinine <=1.5*upper limit of normal (ULN) or calculated creatinine clearance >=50 milliliters per minute (mL/min) using Cockcroft-Gault equation.
  5. Total bilirubin <=1.5*ULN except in participants with Gilbert's syndrome. Participants with Gilbert's syndrome may enroll if direct bilirubin <=1.5*ULN of the direct bilirubin.
  6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.5*ULN.
* Participants must have recovered to Grade 1 toxicity from prior cancer therapy (a participant with Grade 2 neuropathy or Grade 2 alopecia is an exception to this criterion and may qualify for this study).
* Participant able to take oral medications.
* Participant meets the following criteria:

  1. Female participant (of childbearing potential) is not breastfeeding, has a negative serum pregnancy test within 72 hours prior to taking study drug, and agrees to abstain from activities that could result in pregnancy from Screening through 180 days after the last dose of study drug, or is of non-childbearing potential.
  2. Female participant is of non-childbearing potential (other than medical reasons) as defined:

  i) >=45 years of age and has not had menses for >1 year. ii) Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon the screening evaluation.

iii) Has undergone post hysterectomy, bilateral oophorectomy, or tubal ligation. Documented hysterectomy, oophorectomy or tubal ligation must be confirmed in the medical records, otherwise the participant must be willing to use 2 adequate barrier methods throughout the study starting from the screening visit through 180 days after the last dose of study drug. Information must be captured appropriately within the site's source documents.

c) Male participant agrees to use an effective method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

* Able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

* Prior anti-cancer therapies for current malignancy.
* Known evidence of distant metastasis. Staging studies are not required. The decision to pursue staging studies is at the discretion of the treating clinician, based on the participant's clinical and pathological findings consistent with standard guidelines.
* Known hypersensitivity to the components of niraparib components or their formulation excipients.
* Major surgery within 3 weeks of starting the study or participant has not recovered from any effects of any major surgery.
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, uncontrolled hypertension, active uncontrolled coagulopathy, bleeding disorder, or any psychiatric disorder that prohibits obtaining informed consent.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study drug, or is not in the best interest of the participant to participate.
* Participant is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study drug or within the 180-day period after the last dose of study drug.
* Immunocompromised participants.
* Known active hepatic disease (Hepatitis B or C).
* Prior treatment with a known PARP inhibitor.
* Other active malignancy that warrants systemic therapy.
* Known history of myelodysplastic syndromes (MDS) or Acute myeloid leukemia (AML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Spring LM, Han H, Liu MC, Hamilton E, Irie H, Santa-Maria CA, Reeves J, Pan P, Shan M, Tang Y, Graham JR, Hazard S, Ellisen LW, Isakoff SJ. Neoadjuvant study of niraparib in patients with HER2-negative, BRCA-mutated, resectable breast cancer. Nat Cancer. 2022 Aug;3(8):927-931. doi: 10.1038/s43018-022-00400-2. Epub 2022 Jul 4. PMID 35788722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, single-arm pilot study that evaluated the antitumor activity and safety of niraparib as neoadjuvant therapy in participants with human epidermal growth factor receptor 2 (HER2)-negative and breast cancer susceptibility gene mutant (BRCAmut) localized breast cancer.
Pre-assignment Details: A total of 21 participants were enrolled in the study.
Groups:
- Niraparib 200 mg: Participants received niraparib 200 milligrams (mg) orally once daily in 28-day treatment cycles. After 2 cycles, participants either underwent surgery, received additional cycles of niraparib (maximum of 6 cycles total), or received neoadjuvant chemotherapy, at physician's discretion. A breast magnetic resonance imaging (MRI) was performed at the end of cycle 2 and breast ultrasounds were performed at the end of each cycle, including any additional cycles beyond cycle 2. After completion of all neoadjuvant therapy participants proceeded to surgery, at which time pathological complete response (pCR) was assessed.
Period: Overall Study
Arm/Group | Niraparib 200 mg
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Niraparib 200 mg
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Population.
  Years | 44.1 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: Asian | 1
  Race customized: Black or African American | 1
  Race customized: White | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Tumor Response Measured by Breast MRI
Description: Tumor response measured by breast MRI is defined as >=30 percent (%) reduction of tumor volume from Baseline based on primary lesion after niraparib treatment without any new lesion development. Tumor volume was calculated as (length × width × height × pi [π])/6. Responses were assessed as Clinical complete response (CR): A complete disappearance of all tumor signs in the breast as assessed by imaging test. Clinical partial response (PR): A reduction in the tumor volume of the primary tumor size by >=30% assessed by palpation or imaging test. Clinical stable disease (SD): No significant change in tumor volume during treatment. Clinical progressive disease (cPD): The development of new, previously undetected lesions, or an estimated increase in the size of the primary lesion by greater than 20%. Percentage of participants with tumor response and its 95 percent confidence interval (CI) has been presented. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: At 2 months
Population: Efficacy Evaluable Population. The efficacy evaluable population consisted of all participants who completed 2 cycles of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib 200 mg
Number analyzed (Participants) | 21
Percentage of participants | 90.5 [69.6 to 98.8]

2. Secondary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: pCR is defined as ypT0/Tis ypN0 by receipt of pre-operative chemotherapy (Yes versus No). Following neoadjuvant therapy, pathological staging is recorded using the 'yp' designation. ypT0/Tis ypN0 is the absence of invasive cancer in the breast and axillary nodes. pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current American Joint Committee on Cancer [AJCC] staging system). Percentage of participants with pCR rate its 95 percent CI has been presented. CI was based on binomial exact CI.
Time Frame: Up to 1 year
Population: Efficacy Evaluable Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib 200 mg
Number analyzed (Participants) | 21
Percentage of participants | 38.1 [18.1 to 61.6]

3. Secondary Outcome: Percentage of Participants With Tumor Response as Measured by Breast Ultrasound
Description: Tumor response rate was based on the change in tumor volume as measured by breast ultrasound; a response was considered >=30 percent reduction of tumor volume from Baseline without any new lesion development. Tumor volume was calculated as (length × width × height × π)/6. Percentage of participants with tumor response and its 95 percent CI has been presented. CI was based on binomial exact CI.
Time Frame: Up to 6 months
Population: Efficacy Evaluable Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib 200 mg
Number analyzed (Participants) | 21
Percentage of participants | 95.2 [76.2 to 99.9]

4. Secondary Outcome: Percent Change From Baseline in Tumor Volume Measured by Ultrasound
Description: Percentage change in tumor volume from Baseline was measured using ultrasound. Baseline was defined as the most recent measurement prior to the first administration of niraparib. Tumor volume was calculated as (length × width × height × π)/6. The percentage reduction in tumor volume was set as 99% if the tumor becomes too small to measure at the post-baseline visit. Percent change from Baseline was defined as greatest change in volume, derived from all available cycles of niraparib (range from cycle 2 to 6) and multiplied by 100.
Time Frame: Baseline and up to 6 months
Population: Efficacy Evaluable Population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Niraparib 200 mg
Number analyzed (Participants) | 21
Percent change | -83.4 (20.45)

5. Secondary Outcome: Percent Change From Baseline in Tumor Volume Measured by MRI
Description: Percentage change in tumor volume from Baseline after 2 months of niraparib treatment was measured using MRI. Baseline was defined as the most recent measurement prior to the first administration of niraparib. Tumor volume was calculated as (length × width × height × π)/6. The percentage reduction in tumor volume was set as 99% if the tumor becomes too small to measure at the post-baseline visit. Percent change from Baseline was defined as value of post Baseline minus Baseline value and multiplied by 100.
Time Frame: Baseline and at 2 months
Population: Efficacy Evaluable Population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Niraparib 200 mg
Number analyzed (Participants) | 21
Percent change | -77.0 (25.14)

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Treatment Discontinuations and Dose Reductions Due to Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or an important medical event. A TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment.
Time Frame: Up to 1 year
Population: Safety Population. Safety Population comprised of participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 200 mg
Number analyzed (Participants) | 21
Participants
  Any TEAE | 21
  Any SAE | 2
  Any TEAEs leading to nirapirib reduction | 4
  Any TEAEs leading to niraparib discontinuation | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: TEAEs and SAEs were collected in the Safety Population which comprised of participants who received at least one dose of study medication.
Arm/Group | Niraparib 200 mg
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 200 mg (N=21)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 200 mg (N=21)
Nausea (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 14
Mucosal inflammation (General disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypermagnesaemia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Insomnia (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Hot flush (Vascular disorders) | 5
Breast cellulitis (Infections and infestations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Menstruation irregular (Reproductive system and breast disorders) | 2
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03329937/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT03329937/SAP_001.pdf